CLINICAL TRIAL: NCT03202953
Title: Comparison of Volume Controlled Ventilation With 1:1 Inspiratory to Expiratory Ratio and Autoflow-volume Controlled Ventilation in Robot-assisted Laparoscopic Radical Prostatectomy With Steep Trendelenburg Position and Pneumoperitoneum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2017-0400
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Robot Assisted Laparoscopic Prostatectomy

STUDY DESIGN:
Intervention Model Description: 1. 1:1 I:E ratio VCV group
  2. autoflow VCV group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants, investicator, outcome assessors will be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1:1 I:E ratio VCV (Group I) (Experimental): volume controlled ventilation with 1:1 inspiratory to expiratory ratio After trendelenburg position, Tidal volume : 8ml/kg, inspiration:expiration ratio = 1:1, FiO2 = 0.5, maintain end tidal CO2 around 40±5 mmHg. Positive end expiratory pressure will not used.
  Interventions: Procedure: ventilation strategy 1
- autoflow VCV (Group A) (Active Comparator): autoflow volume-controlled ventilation After trendelenburg position, Tidal volume : 8ml/kg, inspiration:expiration ratio = 1:2, FiO2 = 0.5, maintain end tidal CO2 around 40±5 mmHg. Positive end expiratory pressure will not used.
  Interventions: Procedure: ventilation strategy 2

INTERVENTIONS:
Procedure: ventilation strategy 1 — In Group I, after trendelenburg position, patients will be applied 1:1 ratio VCV.
  * Tidal volume : 8ml/kg, inspiration:expiration ratio = 1:1, FiO2 = 0.5, maintain end tidal CO2 around 40±5 mmHg. Positive end expiratory pressure will not used.
  Arms: 1:1 I:E ratio VCV (Group I)
Procedure: ventilation strategy 2 — In group A, after trendelenburg position, patients will be applied autoflow VCV.
  - Tidal volume : 8ml/kg, inspiration:expiration ratio = 1:2, FiO2 = 0.5, maintain end tidal CO2 around 40±5 mmHg. Positive end expiratory pressure will not used.
  Arms: autoflow VCV (Group A)

SUMMARY:
The purpose of this study is to compare the 1: 1 I: E ratio VCV and the autoflow VCV in patients undergoing robot assisted laparoscopic prostatectomy

ELIGIBILITY:
Inclusion Criteria:

1. adult (20-80 years old)
2. patients undergoing robot assisted laparoscopic prostatectomy

Exclusion Criteria:

1. history of COPD
2. decreased heart function (EF <50%)
3. BMI>30
4. patients who cannot read the consent form (e.g., blind, foreigner)

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients undergoing robot assisted laparoscopic prostatectomy
Enrollment: 78 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
PaO2 | 30 minutes after trendelenburg position
  PaO2 analyzed by arterial blood gas analysis

SECONDARY OUTCOMES:
PaO2 | 10 minutes after induction (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3), 10 minutes after supine position (T4)
End tidal CO2 | 10 minutes after induction (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3), 10 minutes after supine position (T4)
peak airway pressure | 10 minutes after induction (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3), 10 minutes after supine position (T4)
blood pressure | 10 minutes after induction (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3), 10 minutes after supine position (T4)
Arterial blood gas analysis | 10 minutes after induction (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3), 10 minutes after supine position (T4)
  pH, SaO2, Base excess

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No